CLINICAL TRIAL: NCT05461638
Title: A Prospective, Randomized, Single-Blinded, Multi-Center, Clinical Trial Comparing Kinematic Alignment vs. Mechanical Alignment Using Medially-Stabilized Knee (GMK Sphere) And Patient-Specific Cutting Guides (MyKnee) For Total Knee Arthroplasty
Brief Title: Kinematic Alignment vs Mechanical Alignment for Total Knee Arthroplasty
Acronym: KA vs MA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No viable sites
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUSA-K-KA-001
Record Dates: First submitted 2022-03-30; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unrestricted Kinematic Alignment (Active Comparator): Mechanical Alignment and Unrestricted Kinematic Alignment using Medacta GMK Sphere with custom cutting guides
  Interventions: Procedure: Mechanical Alignment and Unrestricted Kinematic Alignment using Medacta GMK Sphere with MyKnee Custom guides
- Restricted Kinematic Alignment (Active Comparator): Mechanical Alignment and restricted Kinematic Alignment using Medacta GMK Sphere with custom cutting guides
  Interventions: Procedure: Mechanical Alignment and Restricted Kinematic Alignment using Medacta GMK Sphere with custom cutting guides

INTERVENTIONS:
Procedure: Mechanical Alignment and Unrestricted Kinematic Alignment using Medacta GMK Sphere with MyKnee Custom guides — MA places the implant in an average position for all patients based on pre-determined definition of acceptable knee alignment and has become the most common surgical approach for TKA and Unrestricted KA places the implant in a custom position for each patient, completely matching individual anatomy and restoring natural alignment to that of the prearthritic knee.
  Arms: Unrestricted Kinematic Alignment
Procedure: Mechanical Alignment and Restricted Kinematic Alignment using Medacta GMK Sphere with custom cutting guides — MA places the implant in an average position for all patients based on pre-determined definition of acceptable knee alignment and has become the most common surgical approach for TKA and Restricted KA places the implant in a custom position for each patient, closely matching with anatomy and natural alignment of the individual's knee.
  Arms: Restricted Kinematic Alignment

SUMMARY:
This is a prospective, randomized, single-blinded, multi-center trial comparing Kinematic Alignment vs Mechanical Alignment in TKA patients using patient reported outcomes, clinical and functional performance tests and radiographic analyses.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blinded, multi-center trial comparing Kinematic Alignment vs Mechanical Alignment in TKA patients with Medacta GMK Sphere knee system using patient specific instrumentation Medacta MyKnee. Patients will be assessed a pre-operative, operative and interim post-operative visits, week 6, month 6 and 1,2,5 & 10 years. There will be a phone survey follow up at year 3,4,6,7,8,& 9.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read, understand and provide written informed consent on the Institutional Review Board (IRB) approved Informed Consent Form (ICF).

  * Ability to understand and provide written authorization for use and disclosure of personal health information.
  * Subject who are able and willing to comply with the study protocol and follow-up visits.
  * Must be 21 years or older to participate, and less than 80 years old.
  * Subjects must have osteoarthritis knee disease in the affected knee compliant with the FDA-approved indications for use of GMK Sphere knee system and MyKnee cutting blocks.
  * Patients who are candidates for Total Knee Arthroplasty and are determined to undergo a TKA using the Medacta GMK Sphere implant and MyKnee cutting blocks will be offered enrollment.
  * Subjects must be able to return for the follow-up appointments, and have the mental capacity to cooperate and complete PRO questionnaires, physical exam and radiographs.

Exclusion Criteria:

* • Cases of extreme bone loss requiring an augmented femoral or tibial implant and chronic ligamentous laxity requiring a constrained implant

  * The patient has a fixed flexion deformity of ≥15°
  * The patient has less than 90° of flexion
  * Patient is morbidly obese (BMI ≥40)
  * Patient with inflammatory arthritis
  * History of prior deep knee infection
  * History of alcoholism or drug abuse
  * Currently on chemotherapy or radiation therapy for neoplastic disease
  * Patient currently on immunosuppressive medications including steroids except when, (a) steroid use is less than 10mg daily, (b) other immunosuppressive medications are held for appropriate time, for example Adalimumab is held 2 weeks prior and 2 weeks after surgery
  * History of known sensitivity or allergy to materials used in orthopedic implants, specifically Titanium and Cobalt-Chrome alloys
  * Habitual use of narcotic pain medications prior to surgery (more than 2 doses daily and chronic use of a minimum 3 months)
  * History of metabolic disorder affecting the skeletal system other than osteoarthritis or osteoporosis (e.g., Osteomalacia, Ricketts)
  * History of chronic pain issues for reasons other than knee joint pain. If the type of pain affects activities of daily living, do not enroll. If the pain is intermittent and does not affect activities of daily living, it is OK to enroll. Fibromyalgia is exclusionary.
  * Women who are pregnant
  * Patient with unstable psychiatric illness or psychosis is excluded. (Patients with stable anxiety or depression can be enrolled if PI determines that the condition does not adversely affect study outcomes & requirements)
  * Any patient, in the opinion of the investigator, is unable to fully comply with the surgical, rehabilitation, or follow-up aspects of this procedure.
  * Prior surgery on the target knee other than arthroscopy and/or arthroscopically-assisted ligament reconstruction
  * Prior high tibial osteotomy (HTO) or femoral osteotomy
  * Malunion of fracture of a tibia or femur
  * Patient with a neuromuscular or neurosensory deficiency
  * Patient with history of knee fusion in the affected joint

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-05 (Estimated); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Forgotten Joint Score | Post operative 4-132 months
  Assessment of the improvement of joint specific outcomes following knee replacement surgery using the Knee Forgotten Joint Score

SECONDARY OUTCOMES:
Change from baseline in Knee Osteoarthritis Outcome Score (KOOS) | Baseline to Post operative 4-132 months
  Assessment of improvement of activity levels following knee replacement surgery using the KOOS
Change from baseline in Knee Society Score | Baseline to Post operative 4-132 months
  Patient specific patient outcomes scoring
Change from baseline in Knee Society Score | Baseline to Post operative 4-132 months
  Clinical Exam Range of Motion, Stability and Alignment
Change from baseline in PROMIS | Baseline to Post operative 4-132 months
  Pain Intensity, Pain Interference, and physical function scoring
Change in Baseline in Knee Alignment | Baseline to Post operative 4-132 months
  Determined by radiographic analysis measured by angle of degrees
Change from Baseline of Implant Position Fixation | Baseline to Post operative 4-132 months
  Determined by radiographic analysis by measure radio lucent lines in millimeters

OTHER OUTCOMES:
Number of implant failures, implant survival status | Post operative 4-132 months
  Re-operations, revisions, removals, and device related adverse events
Age of patient | Baseline
  Date of birth
Number of male or female patients | Baseline
  Gender description male or female
Demographics | Baseline
  Height in inches, weight in pounds to determine BMI
Occurrence of prior medical and surgical history | Baseline
  Medical and surgical history of patient prior to knee surgery
Pain medication associated with study knee | Baseline to Post operative 4-132 months
  Pain medication and use of narcotics for the study knee
Return to Work/Activity questionnaire | Baseline to Post operative 4-132 months
  Assessment of ability to return to work or other activities following surgery
Anesthetic | day of surgery
  type of anesthesia used during surgery
Estimated Blood Loss | day of surgery
  Volume of blood loss during surgery
Implant demographics | day of surgery
  Implant femoral and tibial size and poly thickness
Type of Surgical Technique | day of surgery
  Mechanical, Restricted Kinematic, Unrestricted Kinematic and tendon release
Length of Surgery | day of surgery
  Time in minutes skin to skin
Length of Hospital Stay | day of surgery
  Length of stay in hours
Tourniquet Time | day of surgery
  Tourniquet time in minutes
Frequency of Facility type used for knee surgery | day of surgery
  Type of facility used for knee surgery
Complications | Baseline to Post operative 4-132 months
  Assess adverse events and Serious Adverse Events
Assisted device usage | Post operative 4-14 months
  Cessation of assisted device usage by date
Pain, Satisfaction, Narcotics and Function expectations | 36-108 months
  Custom Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Rena Mandino, Study Director — Associate Director, Clinical Research Medacta USA